CLINICAL TRIAL: NCT01988649
Title: The Effect of Intranasal Oxytocin on Pain Sensitivity and Threshold: A Randomized, Double Blinded, Crossover Volunteer Study
Brief Title: Oxytocin and Pain Sensitivity and Threshold
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Duplicate Study
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Walega, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STU00086297
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Pain
Keywords: Pain; Oxytocin
MeSH Terms: conditions — Pain | interventions — Oxytocin; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intranasal Oxytocin (Active Comparator): Administration of 32 units of Oxytocin administered intranasally
  Interventions: Drug: Intranasal Oxytocin
- Placebo (saline) (Placebo Comparator): Administration of 4 sprays intranasally of normal saline.
  Interventions: Drug: Placebo (saline)

INTERVENTIONS:
Drug: Intranasal Oxytocin — Administration of intranasal Oxytocin
  Other Names: Oxytocin
  Arms: Intranasal Oxytocin
Drug: Placebo (saline) — Administration of normal saline intranasally.
  Other Names: normal saline
  Arms: Placebo (saline)

SUMMARY:
Oxytocin is neurohypophysial peptide that acts mainly as a neuromodulator in the brain. In addition,oxytocin have an important roles in sexual reproduction , in particular during and after childbirth. It facilitates birth, maternal bonding, and, breastfeeding. Nasal oxytocin has been commonly used to improve breastfeeding in lactating women. A review of safety , side effects and subjective reaction to intranasal oxytocin in human research in 1529 subjects did not review any differences from placebo. The vast majority of basic science studies suggested a large effect of oxytocin in minimizing acute pain.4 Few studies have demonstrated an association between plasma levels of oxytocin and pain in humans. No studies have examined the effect of intranasal oxytocin on pain sensitivity and threshold. Since addictive properties of oxytocin have not been described, the drug may have important application in the management of acute and chronic pain.

The main objective of the current investigation was to evaluate the effect of intranasal oxytocin on pain sensitivity and threshold in human volunteers. We hypothesized that intranasal oxytocin, in human volunteers ,would decrease sensitivity and and increase pain threshold compared to intranasal saline .

Significance: Intranasal oxytocin may become a viable treatment for acute and chronic pain in humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females volunteers
* English speaking
* Age <20 and > 35

Exclusion Criteria:

* Pregnancy
* Lactation
* Allergy to preservatives
* Mental disease
* Chronic pain
* Current use of analgesics
* Anxiety or depression Drop Out: volunteer request

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Pain sensitivity and threshold | 120 minutes
  Pain sensitivity and threshold using the MEDoc device. Mechanical and thermal pain test will be performed at baseline, before drug administration, at 45 minutes and at 90 minutes.

SECONDARY OUTCOMES:
Side effects of Oxytocin | 2 Hours
  Side effects including running nose, nasal irritation, tears in the eyes.

CONTACTS AND LOCATIONS:
Overall Officials: David Walega, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Yamasue H, Yee JR, Hurlemann R, Rilling JK, Chen FS, Meyer-Lindenberg A, Tost H. Integrative approaches utilizing oxytocin to enhance prosocial behavior: from animal and human social behavior to autistic social dysfunction. J Neurosci. 2012 Oct 10;32(41):14109-17. doi: 10.1523/JNEUROSCI.3327-12.2012. PMID 23055480